CLINICAL TRIAL: NCT06444698
Title: The Effect of Consuming Quinoa on Muscle Strength, VO2max and Athletic Performance Among Adolescent Handball Players
Brief Title: The Effect of Quinoa on Strength, VO2max and Athletic Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Shibili Nuhmani, Assistant Professor, Imam Abdulrahman Bin Faisal University
Allocation: Not Applicable | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-PGS-2023-03-340
Record Dates: First submitted 2024-05-23; First posted 2024-06-05 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-07

CONDITIONS: Sports Nutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): the experimental group will receive two cookies that contain 50 grams of quinoa
  Interventions: Dietary Supplement: cookies that contain 50 grams of quinoa
- Control group (Placebo Comparator): control group will receive the same two cookies that but without quinoa
  Interventions: Dietary Supplement: cookies without quinoa

INTERVENTIONS:
Dietary Supplement: cookies that contain 50 grams of quinoa — 250 grams of ground quinoa will be mixed with 250 grams of ready-to-use cookie flour and 100 gram of butter, one egg, and 75 gram of chocolate chips will be added. After mixing, the ingredients will be divided into (10) cookies (each cookie will continue 25 grams of quinoa) and bake them in oven for 9-11 mint at 190 °C. The placebo control group will receive cookies that continue the same ingredient but without quinoa and the cookies will look like the experimental group cookies. Cookies delivery will be every 3 to 4 days for each participants.
  Arms: Experimental group
Dietary Supplement: cookies without quinoa — The placebo control group will receive cookies that continue the same ingredient of experimental group but without quinoa and the cookies will look like the experimental group cookies.
  Arms: Control group

SUMMARY:
Background: Proper nutrition is essential for sports performance. Quinoa is a gluten-free grain rich in macronutrients such as protein, polysaccharides, and fatty acids and consists of many phytochemicals such as carotenoids, flavonoids, saponins, fiber, vitamins, and minerals. Phytochemicals in quinoa act as antioxidant and anti-inflammatory. This will protect against several oxidative stress related diseases.

Objective: Investigate the effect of 50 g of quinoa for four weeks on muscle strength, VO2max and athletic performance among adolescent athletes.

Study design: A Double blinded randomized control trial with pre-test and post-test design.

Methods :32 subjects will be included in this trial. Subjects will be divided randomly into control and experimental group with a 1:1 ratio; the experimental group will receive two cookies that contain 50 grams of quinoa; the control group will receive the same two cookies that but without quinoa. Strength will be assessed by using hand-held dynamometer (HHD). Maximum oxygen uptake capacity (Vo2max) will be assessed by Queen's College step test (QCT). And for evaluating performance: standing long jump test, ball throw test, and agility T-test will be used. Subjects will be asked to take the cookies 1-4 hours before bedtime daily during the study period.

Statistical Analysis: Shapiro wilk test will be performed to check the normality of the data and Levenes test will be performed to check homogeneity of variance. Cohen's d will be used to check the effect size. The level of significance is set to p ≤ 0.05.

ELIGIBILITY:
Inclusion criteria:

1- Healthy adolescent male athletes aged 15 to 18

Exclusion criteria:

1- Use any dietary supplementation, including protein powder, during the study period.

2. Musculoskeletal, neurological, cardiovascular, or systemic disorders which may affect the testing as reported by the participants

3. Biomechanical abnormalities which may affect the testing as reported by the participants

4. Participants psychological disorders

5. Participants on medication which may affect the measurements as reported by the participants

6. Allergic from any recipe ingredients

Ages: 15 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
strength of the biceps and triceps by Hand held dynameter | base line measurement and post test after 4 weeks of intervention
Maximum oxygen uptake capacity (Vo2max) assessed by Queen's College Step Test (QCT) | base line measurement and post test after 4 weeks of intervention
standing long jump test | base line measurement and post test after 4 weeks of intervention
Ball throw test | base line measurement and post test after 4 weeks of intervention
Agility T-test | base line measurement and post test after 4 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Shibili Nuhmani, PhD, Principal Investigator — Imam Abdulrahman Bin Faisal University
Locations (1):
- Imam abdulrahman bin faisal university, Dammam, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No